CLINICAL TRIAL: NCT04850404
Title: Effect of the Sheath of Rectus Abdominis Block Combined With the Transverse Plane Block on the Condition in Laparoscopic Gynecological Surgery.
Brief Title: Effect of the Sheath of Rectus Abdominis Block Combined With the Transverse Plane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zhangyi, Chief Physician, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1900026767
Record Dates: First submitted 2021-03-25; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Nerve Block; Surgical Conditions
Keywords: TAPB; Moderate NMB; Surgical conditions
MeSH Terms: interventions — Rocuronium; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the group of abdominal nerve block combined with moderate NMB (Experimental): The patients of group N-M received the rectus abdominis block combined with transverse plane block.
  Interventions: Procedure: abdominal nerve block
- moderate NMB group (No Intervention): The patients of group M received moderate NMB through the surgery.

INTERVENTIONS:
Procedure: abdominal nerve block — All Patients of group A-M will be administered with rectus abdominis block combined with TAPB after anesthesia. Rocuronium was infused continuously (concentration: 1 mg/ml) when TOF recovered to 1. The starting rate was 0.3mg/kg/h, and the TOF count was maintained between 1~3 (moderate NMB) and recorded during the operation. Whether and how to add rocuronium was based on TOF count and request of surgeons. When TOF Watch- SX showed 4 or ratio, the investigators increased the speed of rocuronium pump infusion and record the score at the time of shallow NMB. When the chief surgeon thought the vision could not satisfy the needs of the operation, rocuronium 0.1mg/kg in bolus was added as a rescue. Then, the pump speed was lowered or even decreased to 0 to make the TOF count recover to 1~3 as soon as possible.
  Other Names: moderate NMB monitorted by the TOF Watch- SX; Rocuronium; 40 ml of 0.5% ropivacaine
  Arms: the group of abdominal nerve block combined with moderate NMB

SUMMARY:
The situation of demand for surgical conditions is quite high when lymph node resection involved in the surgery type, especially abdominal aortic lymph node dissection, and commonly, the surgeons complained about the interference from the intestine which pushed the investigators to increase the level of neuromuscular blockade close to deep NMB. To avoid the application of deep NMB and promote good surgical conditions for laparoscopic gynecological surgery with lymph nodes resection, the investigators explored other preoperative ways to cooperate with surgeons more harmoniously. It's well known that epidural anesthesia and epidural anesthesia combined with spinal anesthesia have the effect of muscle relaxation which has been applied in clinical practice widely. One study indicated that the Transverse Abdominal Plane (TAP) block could change muscle thickness and achieve the effect of muscle relaxation. It leads investigators to a hypothesis that the sheath of rectus abdominis block combined with transverse abdominal plane block may suppress the signal transmission of abdominal nerve, and may be beneficial to improve surgical conditions.

DETAILED DESCRIPTION:
The investigators conducted this study to test the hypothesis that compared with moderate NMB， the sheath of rectus abdominis block combined with transverse abdominal plane block may reduce the frequency of additional ask for muscle relaxants to optimize surgical conditions, and also provide postoperative analgesia on the premise of moderate NMB.

ELIGIBILITY:
Inclusion Criteria:

1. ASA grade I~ II;
2. aged 18-55 years;
3. BMI 19 ~ 23kg/m2;
4. laparoscopic total hysterectomy and bilateral adnexectomy and/or pelvic lymphadenectomy under elective general anesthesia lasted for more than 2 hours; 5. informed consent has been signed.

Exclusion Criteria:

1. the patient had a history of abdominal surgery;
2. For patients who are professional athletes and weight trainers, abdominal muscle tension can be changed through strength training need to be excluded.
3. allergic to any of the drugs used in the experiment;
4. pregnant or lactating women;
5. patients with severe mental and neurological symptoms cannot cooperate with the study;
6. those who participated in other clinical trials within 3 months before being enrolled in the study;
7. the researcher believes that other reasons are not suitable for clinical trials;
8. patients who have changed their surgical methods or received only palliative surgical treatment;
9. patients with abnormal coagulation function;

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-07-31 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-08-10 (Estimated)

PRIMARY OUTCOMES:
the good or optimal percentage of each group based on the surgical rating scale (5-point scale) | The field of vision was assessed every 15 minutes, from the beginning of the pneumoperitoneum to the end of the pneumoperitoneum. The surgeon gave a score, and the field of vision grade was determined based on the mean value.
  The primary outcome was the frequency of the good or optimal rating scale based on a ﬁve-point surgical rating scale (SRS) ranging from 1 (extremely poor conditions) to 5 (optimal conditions).

IPD SHARING:
Plan to Share IPD: No